CLINICAL TRIAL: NCT05079867
Title: Cochlear Trauma, Functional and Structural Preservation in Cochlear Implant Surgery: Comparative Study Between Perimodiolar and Lateral Wall Electrodes
Brief Title: Cochlear Trauma, Functional and Structural Preservation in Cochlear Implant Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, FEDERICO ALBERTO DI LELLA, MD PhD, Hospital Italiano de Buenos Aires
Other Study IDs: 5906
Record Dates: First submitted 2021-10-03; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss; Cochlear Implant; Cochlear Microphonics; Electrocochleography
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perimodiolar (PM): Patients to be implanted with: Mid Scala or CI532 / 632 (Slim modiolar) electrode
  Interventions: Device: Cochlear implantation
- Lateral wall (PL): Patients to be implanted with: Slim J or CI522 / 622 (Slim Lateral) electrode
  Interventions: Device: Cochlear implantation

INTERVENTIONS:
Device: Cochlear implantation — Electrode surgically implanted in patient's cochlea to improve hearing

SUMMARY:
Prospective 2-arm cohort consisting of a preoperative visit and visits at the time of implantation (Day 0) and follow-up in patients for whom their treating physician indicated a perimodiolar or straight cochlear implant.

DETAILED DESCRIPTION:
Branches:

* Perimodiolar (PM)
* Lateral wall (PL)

Follow up schedule:

Preoperative visit POV1 (up to 90 days before D0) Intraoperative visit D0 (Surgery - Day 0) Follow-up visit 1 FUV1 (48 hours) Follow-up visit 2 FUV2 14 days Follow-up visit 3 FUV3 (4 weeks) Follow-up visit 4 FUV4 (3 months) Follow-up visit 5 FUV5 (6 months) Follow-up visit 6 FUV6 (12 months)

ELIGIBILITY:
Inclusion Criteria:

Patients to receive a Cochlear implant 12 Months of age or older at the time of incorporation Willingness to participate and comply with the requirements of the protocol Residual hearing better than 80 dBA at 500 Hz

Exclusion Criteria:

Medical or pharmacological comorbid condition that contraindicates cochlear implantation.

Previous implantation in the ear of the new implant Ossification or any other cochlear abnormality that could prevent the complete insertion of the electrode guide Abnormal cochlear / neural anatomy on preoperative CT or MRI (excluding dilated vestibular aqueduct syndrome) Deafness due to lesions of the central auditory pathway. (Exclusion for evaluation of residual hearing) Diagnosis of Auditory Neuropathy Spectrum Disorder (Exclusion for evaluation of residual hearing) Active infection in the middle ear Chronic inflammatory processes in the middle ear Disabilities that could prevent participation in the evaluations Unrealistic expectations on the part of the participant regarding the possible benefits, risks and limitations inherent to the procedure or research protocol.

Surgical impossibility to follow the guidelines of the minimally traumatic technique.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients over 12 months of age who will receive a cochlear implant
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-12-19 (Estimated); Study Completion 2023-12-19 (Estimated)

PRIMARY OUTCOMES:
Amplitude of cochlear microphonics | 0-12 months
  Postoperative amplitude of cochlear microphonics

SECONDARY OUTCOMES:
Cochlear implant impedance | 0-12 months
  Postoperative value of cochlear implant impedance
Residual hearing | 0-12 months
  Average audiometric threshold

CONTACTS AND LOCATIONS:
Overall Officials: Federico A Di Lella, MD PhD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Capital Federal, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD to other researchers.